CLINICAL TRIAL: NCT02828748
Title: The Effect of Cannabinoids on Cytokine Production of Colonic Tissue From IBD Patients
Brief Title: Cytokine Production of Colonic Tissue From IBD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, NAFTALI TIMNA, MD, Meir Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0094 MMC
Record Dates: First submitted 2016-06-13; First posted 2016-07-12 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Inflammatory Bowel Disease
Keywords: cannabinoids; inflammatory bowel disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- active UC (Experimental): patients with clinically active ulcerative colitis undergoing colonoscopy not for study purpose, biopsy will be taken from inflamed and normal mucosa and treated with either cannabinoids or will be used as a control
  Interventions: Other: no intervention in patients treatment, only biopsy taken
- remission UC (Experimental): patients with clinically non active ulcerative colitis undergoing colonoscopy not for study purpose, biopsy will be taken from inflamed and normal mucosa and treated with either cannabinoids or will be used as a control
  Interventions: Other: no intervention in patients treatment, only biopsy taken
- active CD (Experimental): patients with clinically active crohns disease undergoing colonoscopy not for study purpose, biopsy will be taken from inflamed and normal mucosa and treated with either cannabinoids or will be used as a control
  Interventions: Other: no intervention in patients treatment, only biopsy taken
- remission CD (Experimental): patients with clinically non active crohns disease undergoing colonoscopy not for study purpose, biopsy will be taken from inflamed and normal mucosa and treated with either cannabinoids or will be used as a control
  Interventions: Other: no intervention in patients treatment, only biopsy taken

INTERVENTIONS:
Other: no intervention in patients treatment, only biopsy taken

SUMMARY:
Chronic intestinal inflammation characterizes inflammatory bowel diseases (IBD), which consist mainly of Crohn's disease and ulcerative colitis. The exact etiology is unknown for both diseases and therapeutic attempts aimed at down-regulating intestinal inflammation use both mediator-specific and nonspecific immune suppression. These attempts cause considerable side effects. Also, IBD patients are different in their genetic background and pathology. It was previously shown that products based on marijuana (Cannabis sativa) produce beneficial effects for patients with IBD, and medical cannabis-based products were formerly proven to have anti-inflammatory activity in laboratory experiments and in clinical tests. However, it is unknown how C. sativa-based medical products exert their effect in IBD and additional research and development should be done. One issue to be resolved in the process of medicalization of C. sativa is the base for the differences in patient response to different C. sativa lines, in order to fine-tune C. sativa -based treatment to IBD patients.

For this aim of fine-tuning C. sativa -based treatment to IBD patients, we characterized the chemical composition of different C. sativa lines and their anti-inflammatory activities on colon cells lines. Extracts of C. sativa lines were prepared using various methods and cannabinoids and terpenoids profile was determined by chemical analysis. We found that different compounds have different effects on inflamed colon cell lines, leading to changes in interleukin secretion, inflammation markers and gene expression in the treated colon cells. In addition, we have developed a unique system relevant for personalized medicine in IBD. This system allows a patient-specific determination of the effect of C. sativa -based treatment. Following, clinical tests will be conducted aiming to develop cannabis-based products from different C. sativa lines, with anti-inflammatory activity that is effective and optimized for the different IBD patients.

DETAILED DESCRIPTION:
Title of the project:

Efficacy of cannabinoids in the treatment of inflammatory bowel disease

Question to be investigated:

The marijuana plant, Cannabis sativa has been used as a medicinal treatment for a variety of diseases. Cannabinoids have been reported to alleviate neurological conditions including MS-related symptoms such as spasticity, pain, tremor and bladder dysfunction . Other neurological conditions, such as chronic intractable pain, dystonic movement disorders, and Tourette's Syndrome were also reported to be alleviated by cannabis use . Cannabis has been used to treat anorexia in AIDS and cancer patients. In gastroenterology, cannabis has been used to treat anorexia, emesis, abdominal pain, gastroenteritis, diarrhea, intestinal inflammation, and diabetic gastroparesis .

The cannabis plant contains over 60 different compounds which are collectively referred to as cannabinoids . Of these, the two compounds delta 9-tetrahydrocannabinol (THC) and Cannabidiol (CBD) seem to be the most active.

Cannabinoids have a profound anti-inflammatory effect, mainly through the CB2 receptor. Cell mediated immunity was found to be impaired in chronic marijuana users . A potent anti-inflammatory effect of cannabis was observed in rodents. Studying the functional roles of the endocannabinoid system in immune modulation reveals that it is involved in almost all major immune events. Cannabinoids shift the balance of pro-inflammatory cytokines and anti-inflammatory cytokines towards the T-helper cell type 2 profiles (Th2 phenotype) and suppress cell-mediated immunity, whereas humoral immunity may be enhanced. Cannabidiol was shown to reduce inflammation in a mouse model of rheumatoid arthritis and type I diabetes mellitus.

Therefore, cannabinoids can be used to treat various inflammatory conditions including rheumatoid arthritis and asthma.

In the gut, Endocannabinoids are produced by both the serosal and mucosal component of the human intestine, and studies on cell lines have shown that human intestinal epithelial cells can produce endocannabinoids; additional sources of endocannabinoids in the gut include human endothelial cells, platelets, resident macrophages and other immune cells such as lymphocytes. CB1 and CB2 receptors are be upregulated in experimental models of inflammatory bowel disease. In a mouse model of colitis, cannabinoids were found to ameliorate inflammation, and in the human intestine, levels of Anandamide are increased during inflammation. The inflamed small intestine also has significantly elevated activity of FAAH as well as expression of CB1 cannabinoid receptors.

The exact cellular targets implicated in the reduction of inflammation by cannabinoids are unknown. In a model of bronchopulmonary inflammation in mice administration of anandamide decreased TNF alpha levels in bronchoalveolar lavage fluid. Delta 9-tetrahydrocannabinol (THC) inhibits synthesis of IL-12, IL-2, IL-6, INF gamma, and T cell proliferation.

Many patients with IBD report that smoking marihuana ameliorated their symptoms, but there are no clinical studies investigating that observation. We have recently published the first reported observation of use of medical cannabis in Crohn's disease. In our study, of 30 patients, 21 improved significantly after treatment with cannabis. The average Harvey Bradshaw index improved from 14 ± 6.7 to 7 ± 4.7 (P < 0.001). Number of bowel movements was reduced from an average of eight a day to five a day and the need for other medication, particularly steroids, was significantly reduced. In view of those results we conducted a double blind placebo controlled trial in 20 active Crohn's disease patients. Patients with a Crohn's Disease Activity Index (CDAI)>200 who did not respond to steroids, immunosuppressants or anti-TNF were randomized to receive 2 cigarettes of cannabis or placebo daily. Each cigarette contained 0.5 g of cannabis, corresponding to 11.5mg Tetrahydrocannabinol (THC). The placebo contained cannabis leaves from which THC was extracted. During treatment the CDAI changed in the cannabis group from 358 ± 99 to 139±111 (p<0.05) and in the placebo group from 373 ± 94 to 306±143 (p=Non significant). Five patients in the cannabis group and one in the placebo group went into complete remission (CDAI <100). Three steroid dependent patients in the cannabis group stopped steroids during the study. Patients reported improved appetite and sleep, with no serious side effects.

These preliminary data indicate that cannabinoids have a great potential in the treatment of Crohn's disease, but further investigation of their influence, mode of action, active and non active cannabinoids and alternative routs of application is clearly needed. Most important is the question whether the improvement observed with cannabis consumption is only symptomatic or whether there is a real improvement in inflammation.

The aim of the proposed study is to evaluate inflammation and cytokine levels in explants of colonic tissue from IBD patients with and without cannabidiol.

Materials and methods:

Study population: Patients with either Crohn's disease or ulcerative colitis scheduled for colonoscopy as deemed necessary by their physician will be eligible for the study. After obtaining informed consent, biopsies from inflamed and normal tissue will be taken and processed in a tissue culture media as described further. There will be 6 biopsies from each site.

Methods:

Explants will be cultured in groups of three with the villus surface up on microporous membranes (0.45-_m pore size) contained in Millicell-HA tissue culture inserts (Millipore). The inserts will be placed inside 6-well plastic tissue culture dishes (Costar 3506) along with 1.5 ml of tissue culture medium. Tissue culture medium will be Dulbecco's modified Eagle's medium supplemented with 10% heat-inactivated fetal calf serum, penicillin (100units/ml), streptomycin (100 μg/ml), leupeptin (50 μg/ml), PMSF (1 mM), soybean trypsin inhibitor (50 μg/ml), and dexamethasone (200 μg/ml). Cultures will be incubated at 37°C incubator and gassed hourly with95% oxygen 5% carbon dioxide. Six biopsies from each site will be obtained. Three biopsies will serve as a control and three will be cultured with the addition of Cannabidiol (1 μg/ml). After 24 hours tissue viability will be assessed by addition of Alamar to one of each 3 samples. Change of color from purple to pink indicates viable tissue. The supernatant from the other 4 biopsies will be collected and frozen at -20°C. The biopsies will than be placed in formalin for pathology inspection.

The supernatant from controlled and cannabis treated samples will be analyzed for the presence and level of TNF alpha, Interferon gamma,IL-23, IL-12, IL-2, IL-10, IL-17 and IL-6.

ELIGIBILITY:
Inclusion Criteria:

* established diagnosis if IBD informed consent

Exclusion Criteria:

* contra indication for a biopsy, such as a risk of hemorrhage

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-07 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
reduction of TNF alpha by more them 50% when cannabinoids appllied to culture | 24 hours
  different extracts of cannabis sativa will be applied to culture of biopsy and the cytokins TNF alpha, will be measured in the supernatant of the treated biopsies and compared to controls
reduction of IL-6 by more them 50% when cannabinoids applied to culture | 24 hours
  different extracts of cannabis sativa will be applied to culture of biopsy and the cytokin IL-6, will be measured in pg/ml in the supernatant of the treated biopsies and compared to controls
reduction of IL-8 by more them 50% when cannabinoids applied to culture | 24 hours
  different extracts of cannabis sativa will be applied to culture of biopsy and the cytokine IL-8, will be measured in pg/ml in the supernatant of the treated biopsies and compared to controls
reduction of IL-17 by more them 50% when cannabinoids applied to culture | 24 hours
  different extracts of cannabis sativa will be applied to culture of biopsy and the cytokine IL-17, will be measured in pg/ml in the supernatant of the treated biopsies and compared to controls
increase of IL-10 by more them 50% when cannabinoids applied to culture | 24 hours
  different extracts of cannabis sativa will be applied to culture of biopsy and the cytokine IL-10, will be measured in pg/ml in the supernatant of the treated biopsies and compared to controls

CONTACTS AND LOCATIONS:
Overall Officials: Fred Konnikoff, MD, Study Chair — Meir Medical Center
Locations (1):
- Gastroenterology institute Meir Hospital, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Browning TH, Trier JS. Organ culture of mucosal biopsies of human small intestine. J Clin Invest. 1969 Aug;48(8):1423-32. doi: 10.1172/JCI106108. PMID 5796354
- [Result] Naftali T, Bar-Lev Schleider L, Dotan I, Lansky EP, Sklerovsky Benjaminov F, Konikoff FM. Cannabis induces a clinical response in patients with Crohn's disease: a prospective placebo-controlled study. Clin Gastroenterol Hepatol. 2013 Oct;11(10):1276-1280.e1. doi: 10.1016/j.cgh.2013.04.034. Epub 2013 May 4. PMID 23648372